CLINICAL TRIAL: NCT06732921
Title: Protocol for a Pilot Interventional Study Evaluating the Efficiency and Safety of a Telemedicine Solution for the Post-Anesthesia Care Unit
Brief Title: Recovery Control Tower Feasibility Pilot
Acronym: RCT Pilot
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Michael Avidan, Chair, Department of Anesthesiology, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202305152
Record Dates: First submitted 2023-09-18; First posted 2024-12-13 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Elective Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Recovery Control Tower (RCT) (Experimental): Clinicians in the RCT will remotely work with PACU clinicians to care for patients assigned to one of the two study bays. A version of AlertWatch® (AlertWatch, Ann Arbor, Michigan) decision-support software, customized for the PACU environment, will assist clinicians in the RCT to perform core PACU-related functions remotely. Caregility's iObserver, from the Caregility Cloud™ Virtual Care Platform, will be used for two-way video communication When feasible, RCT clinicians will join handoff activities from the OR to the PACU and discuss pertinent intraoperative events with clinical teams on the ground. RCT clinicians will document patient specific recovery tasks within AlertWatch to assist in tracking patient recovery progresses. RCT clinicians will be the initial point of contact for ongoing recovery care, such as order placements. The attending anesthesiologist in the RCT will assess patients' discharge readiness throughout their PACU stay.
  Interventions: Device: Alertwatch - Recovery Control Tower

INTERVENTIONS:
Device: Alertwatch - Recovery Control Tower — Decision-support software, customized for the PACU environment, Interaction between the telemedicine center and the PACU

SUMMARY:
A pilot study in perioperative telemedicine that aims to demonstrate the efficiency, and safety of integrating telemedicine into the PACU environment. This pilot study will expand on our previously conducted proof-of-concept study for a telemedicine solution in the PACU. If this pilot study proves to be successful, the study team intends subsequently to expand such a telemedicine solution to multiple clinical locations.

ELIGIBILITY:
* Adults (18 years and older)
* Undergoing elective surgery at Barnes Jewish Hospital in St. Louis, Missouri will be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8500 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Time spent in PACU | Day of surgery
  Time patient enters PACU to time patient leaves PACU

SECONDARY OUTCOMES:
Time to PACU sign-out by anesthesia clinician | From the time the patient enters post-anesthesia care unit until time patient leaves post-anesthesia care unit, assessed up to 24 hours after surgery.
  Time patient enters PACU to time discharge note is signed in EHR by anesthesiologist
Pain score in PACU | From the time the patient enters post-anesthesia care unit until time patient leaves post-anesthesia care unit, assessed up to 24 hours after surgery.
  0 to 10 (numeric rating scale [NRS]) - 0 correspond to no pain, ≤ 3 to mild pain, 4-6 to moderate, and scores ≥7 to severe pain
PONV status in PACU | From the time the patient enters post-anesthesia care unit until time patient leaves post-anesthesia care unit, assessed up to 24 hours after surgery.
  None, resolved, resolved and tolerable, persists despite treatment, unable to evaluate
Clinician interactions - Number of contacts RCT clinicians receive from PACU clinicians | From the time the patient enters post-anesthesia care unit until time patient leaves post-anesthesia care unit, assessed up to 24 hours after surgery.
  Reason for contact will be logged (i.e. order placement requests, patient assessments)
Clinician interactions - Number of contacts RCT clinicians make to PACU clinicians for on-the-ground intervention | From the time the patient enters post-anesthesia care unit until time patient leaves post-anesthesia care unit, assessed up to 24 hours after surgery.
  Reason for contact will be logged
Safety events - Return to hospital | 24 hours
  New admission notes, and ED/urgent care notes
Safety events - Number of participants with elevation of care | 24 Hours
  Patients with floor to ICU transfer, and unplanned floor to OR (return to OR)
Safety events - Number of participants with administration of rescue drugs | 24 Hours
  Events of Naloxone (opioid overdose) and Flumazenil (benzodiazepine overdose) administration
Safety events - Significant event notes | 24 Hours
  To identify death events
PACU clinician satisfaction | Through study completion, an average of 1 year
  From monthly surveys

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Avidan, MBBcH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No